CLINICAL TRIAL: NCT01146795
Title: Feasibility of Carboplatin, Paclitaxel and Bevacizumab Neoadjuvant Therapy for Epithelial Ovarian, Fallopian Tube and Primary Peritoneal Cancer
Brief Title: Neoadjuvant Therapy for Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jason D. Wright (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jason D. Wright, Sol Goldman Associate Professor of Gynecology Oncology (in Obstetrics and Gynecology), Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAD8429
Record Dates: First submitted 2010-05-21; First posted 2010-06-22 (Estimated); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal Cancer; Fallopian Tube Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carboplatin, Paclitaxel, and Bevacizumab (Experimental): Three 21 day cycles of carboplatin, paclitaxel, and bevacizumab.
  After 3 cycles of chemotherapy patients will be considered for surgical cytoreduction. Patients must fulfill all criteria to be considered eligible for surgical exploration: 1) ≥50% reduction in pretreatment cancer antigen 125 (CA-125) and 2) No medical contraindications to surgery.
  After surgical cytoreduction all patients will receive an additional 6 cycles of chemotherapy (cycles 4-9) regardless of disease status at the time of exploration. Chemotherapy should be re-instituted within 6 weeks of the surgical procedure. Bevacizumab will be omitted from cycle 4 of chemotherapy. Patients who do NOT undergo surgical resection should receive cycles 4-9 of therapy. In this instance bevacizumab may be included in cycle 4.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be administered at a concentration-time curve (AUC) of 5-6 (at the discretion of the physician) day 1 every 3 weeks in combination with Paclitaxel and Bevacizumab.
  Other Names: Paraplatin
Drug: Paclitaxel — Paclitaxel 175 mg/m2 over 3 hours day 1 every 3 weeks in combination with Carboplatin and Bevacizumab.
  Other Names: Taxol
Drug: Bevacizumab — Bevacizumab 15 mg/kg day 1 every 3 weeks in combination with Paclitaxel and Carboplatin.
  Other Names: Avastin

SUMMARY:
This study is to determine the feasibility of administering neoadjuvant carboplatin, paclitaxel, and bevacizumab without excessive dose modification or cycle delay in patients with epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer. This study will also investigate the rate of optimal cytoreduction, response rate and progression free and overall survival, and to assess the quality of life for patients with epithelial ovarian cancer, primary peritoneal cancer or fallopian tube cancer treated with neoadjuvant carboplatin, paclitaxel and bevacizumab.

DETAILED DESCRIPTION:
Initial treatment for ovarian cancer is usually surgical cytoreduction followed by adjuvant platinum and taxane chemotherapy. At the time of diagnosis over 75% of patients present with stage III or IV disease that has spread into the peritoneal cavity or distally. Despite a number of new chemotherapeutic regimens survival has improved only modestly over the preceding two decades. While overall 5-year survival has improved from 30% to 50%, 5-year survival remains only 25% for women with advanced stage disease. Given these findings it is clear that improved strategies for the delivery of cytotoxic and biologic agents are needed for women with advanced stage epithelial ovarian cancer.

A newer drug, called bevacizumab, has been approved by the U.S. Food and Drug Administration (FDA) for use in combination with chemotherapy in patients with colon cancer, lung cancer, and some types of breast cancer that have spread to distant sites in the body. A critical question which will need to be answered is whether or not it is feasible to administer a combination of bevacizumab with standard cytotoxic therapy using a neo-adjuvant approach for patients with epithelial cancer of the ovary, fallopian tube, or primary peritoneum.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have Suspected Federation of Gynecology and Obstetrics (FIGO) stage III or IV disease.
* Cytologic or histologic diagnosis of a carcinoma felt by the investigator to be compatible with epithelial cancer of the ovary, fallopian tube, or primary peritoneum
* Patients must have a Performance Status of 0, 1 or 2.
* Patients with prior anthracycline exposure must have a baseline multigated acquisition scan (MUGA) or echocardiogram prior to study entry.
* Patients must have adequate:

  * Bone marrow function: Absolute neutrophil count (ANC) greater than or equal to 1500/υl, equivalent to Common Toxicity Criteria for Adverse Events v3.0 (CTCAE) Grade 1. This ANC cannot have been induced or supported by granulocyte colony stimulating factors.
  * Platelets greater than or equal to 100,000/υl (CTCAE Grade 0-1).
  * Hematocrit > 21%.
  * Renal function: Creatinine < 1.5 x institutional upper limit of normal (ULN), CTCAE Grade 1.
  * Hepatic function: Bilirubin less than or equal to 1.5 x ULN (CTCAE Grade 1). AST, ALT, and alkaline phosphatase less than or equal to 2.5 x ULN (CTCAE Grade 1). Aspartate transaminase (AST) and alanine transaminase (ALT)
  * Neurologic function: Neuropathy (sensory and motor) less than or equal to CTCAE Grade 1.
  * Coagulation function: Prothrombin Time (PT) and Partial Thromboplastin Time (PTT) - PT such that international normalized ratio (INR) is ≤ 1.5 (or an in-range INR, usually between 2 and 3, if a patient is on a stable dose of therapeutic warfarin for management of venous thrombosis including pulmonary thromboembolism) and a PTT < 1.2 times the upper limit of normal.
* Patients must have measurable disease. Patients may or may not have cancer-related symptoms.
* Baseline CA-125 must be ≥ 70 units/mL.
* Patients must have met all pre-entry requirements.
* An approved informed consent and authorization permitting release of personal health information must be signed by the patient or guardian.
* Eligible patients should be deemed as likely to be medically fit to undergo surgical cytoreduction after 3 cycles of neoadjuvant chemotherapy by a surgical gynecologic oncologist.
* Patients may receive estrogen +/- progestin replacement.

Exclusion Criteria:

* Patients should NOT have undergone any prior cancer directed surgery (exploration, debulking, etc), with the exception of a minor procedure such as biopsy or cytology specimen.
* Patients who have received prior chemotherapy, immunotherapy, radiotherapy, hormonal therapy or biologic therapy for their ovarian or primary peritoneal cancer are not eligible.
* Patients with borderline ovarian tumors, recurrent epithelial ovarian or primary peritoneal cancer or non-epithelial ovarian cancer are not eligible.
* Patients with a CA125:CEA ratio <25. Carcinoembryonic Antigen (CEA)
* Patients with other cancers (other than non-melanoma skin cancer) within the last five years.
* Patients with acute hepatitis or end stage liver disease.
* Patients with serious non-healing wound, ulcer or bone fracture. This includes history of abdominal fistula or intra-abdominal abscess within 6 months. Patients with granulating incisions healing by secondary intention with no evidence of fascial dehiscence or infection are eligible but require weekly wound examinations.
* History of prior gastrointestinal perforation.
* Patients with evidence of abdominal free air not explained by paracentesis.
* Patients with signs or symptoms of gastrointestinal obstruction including those receiving total parenteral nutrition (TPN), intravenous hydration or tube feeds.
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels by imaging, regardless of whether any chance of requiring vascular reconstruction.
* Patients with history or evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within six months of the first date of treatment on this study. Patients with treated brain metastases can enter the study. Treated brain metastases are defined as having no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period. Anticonvulsants (stable dose) are allowed. Treatment for brain metastases may include whole brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, LINAC, or equivalent) or a combination as deemed appropriate by the treating physician. Patients with central nervous system (CNS) metastases treated by neurosurgical resection or brain biopsy performed within 3 months prior to Day 1 will be excluded.
* Patients with clinically significant cardiovascular disease. This includes:

  * Uncontrolled hypertension, defined as systolic > 140 mm Hg or diastolic > 90 mm Hg.
  * Myocardial infarction or unstable angina within 6 months of day 1 prior to registration.
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure.
  * Serious cardiac arrhythmia requiring medication. This does not include atrial fibrillation.
  * CTCAE Grade 3 or greater peripheral vascular disease.
  * History of CVA within six months.
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies including hypersensitivity to any component of bevacizumab
* Patients with clinically significant proteinuria. Urine protein should be screened by urine protein-creatinine ratio (UPCR). The UPCR has been found to correlate directly with the amount of protein excreted in a 24 hour urine collection. Specifically, a UPCR of 1.0 is equivalent to 1.0 grams of protein in a 24 hour urine collection. Obtain at least 4 ml of a random urine sample in a sterile container (does not have to be a 24 hour urine). Send sample to lab with request for urine protein and creatinine levels (separate requests). The lab will measure protein concentration (mg/dL) and creatinine concentration (mg/dL). The UPCR is derived as follows: protein concentration (mg/dL)/creatinine (mg/dL). Patients must have a UPCR < 1.0 to allow participation in the study.
* Patients with hypertensive crises or hypertensive encephalopathy
* History of hemoptysis (≥ ½ teaspoon of bright red blood per episode) within 1 month prior to day 1.
* Patients with or with anticipation of a non-study related invasive procedure defined as followed:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to the first date of bevacizumab.
  * Major non-study related surgical procedure anticipated during the course of the study.
  * Core biopsy within 7 days prior to first date of bevacizumab.
* Patients with a Performance Status of Grade 3 or 4 are not eligible.
* Patients who are pregnant or nursing. Subjects of child-bearing age have to use effective means of contraception.
* Patients under the age of 18.
* Patients who have received prior therapy with any anti-VEGF drug, including bevacizumab. Vascular endothelial growth factor (VEGF)
* Patients with human immunodeficiency virus (HIV).
* Patients with medical history or conditions not otherwise previously specified which in the opinion of the investigator should exclude participation in this study. The investigator should consult the Study Chair.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-05-17 (Actual); Primary Completion 2015-04-13 (Actual); Study Completion 2015-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Wright, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Columbia University Medical Center, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No significant events in the study that occurred after participant enrollment but prior to assignment of participants to an arm or group.
Groups:
- Carboplatin, Paclitaxel, and Bevacizumab: Three 21 day cycles of carboplatin, paclitaxel, and bevacizumab. After 3 cycles of chemotherapy patients will be considered for surgical cytoreduction. After surgical cytoreduction all patients will receive an additional 6 cycles of chemotherapy (cycles 4-9) regardless of disease status at the time of exploration. Chemotherapy should be re-instituted within 6 weeks of the surgical procedure.
Period: Overall Study
Arm/Group | Carboplatin, Paclitaxel, and Bevacizumab
Started | 32
Completed | 12
Not Completed | 20
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 6
Not completed — Still in treatment at study closure | 10

BASELINE CHARACTERISTICS:
Population: Women with metastatic ovarian, fallopian tube, or primary peritoneal cancer.
Arm/Group | Carboplatin, Paclitaxel, and Bevacizumab
Number analyzed (Participants) | 32
Age, Customized [Count of Participants; unit: Participants]
  Age: 40-49 | 3
  Age: 50-59 | 4
  Age: 60-69 | 13
  Age: 70-79 | 9
  Age: 80-89 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Protocol Defined Adverse Events in Patients Receiving Neoadjuvant Carboplatin, Paclitaxel, and Bevacizumab
Description: This is to assess the feasibility of delivering multiple cycles of the study treatment without excessive dose modification or cycle delays. The regimen would be considered unfeasible for further study if there were 5 or more of the following events within the first 15 patients, 7 or more of these events within the first 30 patients, or 8 or more of these events within the first 45 patients:
  * Delay of day 1 of therapy > 3 weeks from the expected day 1 of that cycle
  * Febrile neutropenia requiring hospitalization
  * Grade 4 thrombocytopenia
  * Grade 1-5 gastrointestinal perforation
  * Grade 3-4 hemorrhagic toxicity
  * Grade 3-4 arterial thromboembolic complications
  * Grade 4 hypertension
  * Grade 4 proteinuria
  * Fascial dehiscence
Time Frame: Up to 30 days after completion of 9 cycles of treatment and/or early discontinuation (approximately up to 12 months)
Population: 32 patients, out of the 45 targeted accrual, were enrolled during the study period. In the first 30 patients, toxicities were analyzed for this outcome measure.
Measure: Number; unit: protocol defined adverse events
Arm/Group | Carboplatin, Paclitaxel, and Bevacizumab
Number analyzed (Participants) | 30
protocol defined adverse events | 7

2. Secondary Outcome: Response Rate
Description: The percentage of patients whose cancer shrinks or disappears after treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Cycle 3, Cycle 6, Cycle 9 and 3 years post-treatment
Population: 31 patients, out of 32 enrolled, were potential candidates for surgery and included in the analysis for this outcome measure. At the time of study, data was only analyzed after 3 cycles of treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Carboplatin, Paclitaxel, and Bevacizumab
Number analyzed (Participants) | 31
percentage of patients
  Complete response | 6.5
  Partial response | 71.0
  Stable disease | 22.6

3. Secondary Outcome: Quality of Life (QOL) Score
Description: The FACT Quality of Life (QOL) Score questionnaire is designed to assess the effects of cancer and its treatment on the quality of life, by measuring aspects of an individual's sense of well-being and ability to carry out various activities. When calculating the total QOL score, the score scale of functional well-being was reversed in order to keep consistent with other three domains. The lower the total score, the better the quality of life. The five-point scale ranges from 0 (not at all) to 4 (very much). Scoring the FACT-G is performed through a simple sum of item scores. Each subscale is scored, and a total score for the FACT-G is obtained by adding each of the subscale scores. With a total possible score greater than 100, additional scoring methods have been used to simplify interpretation. Modifications of scoring include normalizing the total score on a scale of 0-100 through mathematical transformations, as well as the use of a Trial Outcome Index (TOI).
Time Frame: Baseline, Cycle 3, Cycle 6, Cycle 9
Population: A total of 30 patients contributed data to QOL at baseline, not all patients completed the subsequent cycles as demonstrated in the "Number Analyzed" at Cycles 3, 6 and 9.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Carboplatin, Paclitaxel, and Bevacizumab
Number analyzed (Participants) | 30
score on a scale
  Baseline Quality of Life (QOL) Score | 6 (4)
  Cycle 3 Quality of Life (QOL) Score: number analyzed (Participants) | 24
  Cycle 3 Quality of Life (QOL) Score | 7.4 (5.7)
  Cycle 6 Quality of Life (QOL) Score: number analyzed (Participants) | 18
  Cycle 6 Quality of Life (QOL) Score | 8.9 (6.2)
  Cycle 9 Quality of Life (QOL) Score: number analyzed (Participants) | 12
  Cycle 9 Quality of Life (QOL) Score | 6.6 (4.3)

4. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time during and after the treatment of cancer, that a patient lives with the disease but it does not get worse.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin, Paclitaxel, and Bevacizumab
Number analyzed (Participants) | 32
months | 16.8 [12.7 to 20.8]

ADVERSE EVENTS:
Time Frame: Up to 30 days after completion of 9 cycles of treatment and/or early discontinuation (approximately up to 12 months).
Description: Adverse Events Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Carboplatin, Paclitaxel, and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 4/32
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Paclitaxel, and Bevacizumab (N=32)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 — Grade 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin, Paclitaxel, and Bevacizumab (N=32)
Sensory neuropathy (Nervous system disorders) | 29
Motor neuropathy (Nervous system disorders) | 2 — Grade 2
Mood alteration: Anxiety (Nervous system disorders) | 3 — Grade 1
Headache (Nervous system disorders) | 6
Gait Abnormal (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2
Edema, limb (Blood and lymphatic system disorders) | 5
Edema, trunk/genital (Musculoskeletal and connective tissue disorders) | 2
Decreased hemoglobin (Blood and lymphatic system disorders) | 31
Decreased Leukocytes (Blood and lymphatic system disorders) | 26
Decreased ANC (Blood and lymphatic system disorders) | 17 — Grade 1-2
Decreased ANC (Blood and lymphatic system disorders) | 30 — Grade 3-4
Hyponatremia (Blood and lymphatic system disorders) | 11
Hypoglycemia (Blood and lymphatic system disorders) | 3
Hypercalcemia (Blood and lymphatic system disorders) | 3
Hypocalcemia (Blood and lymphatic system disorders) | 7
Hyperglycemia (Blood and lymphatic system disorders) | 17
Hypoalbuminemia (Blood and lymphatic system disorders) | 7
Hyperkalemia (Blood and lymphatic system disorders) | 5
Hypokalemia (Blood and lymphatic system disorders) | 2
Hypomagnesemia (Blood and lymphatic system disorders) | 11
Elevated AST/SGOT (Blood and lymphatic system disorders) | 4
Alkaline phosphatase increased (Blood and lymphatic system disorders) | 3
Hemolysis (Blood and lymphatic system disorders) | 4
INR increased (Blood and lymphatic system disorders) | 4
PTT increased (Blood and lymphatic system disorders) | 3
Decreased platelets (Blood and lymphatic system disorders) | 23
Hemorrhage, nasal (Respiratory, thoracic and mediastinal disorders) | 7
Nausea (Gastrointestinal disorders) | 22
Vomiting (Gastrointestinal disorders) | 6
Taste alteration (Gastrointestinal disorders) | 5
Anorexia (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 14
Flatulence (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 24
Abdominal distension (Gastrointestinal disorders) | 5
Heartburn (Gastrointestinal disorders) | 7
Gastric mucositis (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Fever (General disorders) | 5 — Grade 1
Sweating (General disorders) | 4
Insomnia (General disorders) | 10
Fatigue (General disorders) | 24 — Grade 1-2
Weight loss (General disorders) | 7
Rigors (General disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 4
Flushing skin (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 8 — Grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 20 — Grade 1
Alopecia (Skin and subcutaneous tissue disorders) | 13 — Grade 2
Acne (Skin and subcutaneous tissue disorders) | 3
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Ear, nose and throat exam abnormal (Ear and labyrinth disorders) | 6
Hypertension (Vascular disorders) | 18
Palpitations (Cardiac disorders) | 4
Hot flashes (Vascular disorders) | 3
Rhinitis (Immune system disorders) | 9
Increased creatinine (Renal and urinary disorders) | 5
Proteinuria (Renal and urinary disorders) | 8
Urine incontinence (Renal and urinary disorders) | 3
Wound complication - non-infectious (Surgical and medical procedures) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2 — Grade 1
Abdominal pain (Gastrointestinal disorders) | 9
Joint pain (Gastrointestinal disorders) | 15 — Grade 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 — Grade 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Pain (General disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Febrile neutropenia (Infections and infestations) | 2 — Grade 3
Urinary tract infection (Infections and infestations) | 2 — Grade 2
Infection, other (Infections and infestations) | 2 — Grade 1
Cytokine release syndrome (Immune system disorders) | 2 — Grade 2
Thrombosis (Vascular disorders) | 2 — Grade 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes